CLINICAL TRIAL: NCT05113927
Title: A Prospective, Multi-center, Randomized, Double-arm Trial to Determine the Impact of the SELENE System on Positive Margin Rates in Breast Conservation Surgery.
Brief Title: Wide Field OCT + AI for Positive Margin Rates in Breast Conservation Surgery.
Acronym: RCT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Perimeter Medical Imaging (Industry)
Collaborators: Cancer Prevention Research Institute of Texas (Other); Proxima CRO (Industry); Biostatistical Consulting, Inc. (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: PER-19-04
Record Dates: First submitted 2021-11-02; First posted 2021-11-09 (Actual); Last update posted 2024-12-02 (Actual); Status verified 2024-11

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Intervention Model Description: Multi-center, randomized, double-arm trial
Who Masked: Participant, Care Provider, Investigator
Masking Description: The pathologist at each participating site will be blinded to the study arm to ensure that the pathological assessment is unbiased. Additionally, the subject will be blinded to their randomization until the BREAST-Q questionnaire has been completed.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (2):
- Standard of Care (No Intervention): Lumpectomy with usual intraoperative margin assessment
- Device (Experimental): Imaging of all margins with investigational device
  Interventions: Device: Selene

INTERVENTIONS:
Device: Selene — SELENE imaging of all margins, with record of each margin assessment and an opportunity to excise tissue from the lumpectomy cavity post-imaging. The new margin will be imaged with SELENE and the surgeon will record the assessment and may take additional tissue (up to a maximum of six total shaves, including up to two shaves in each orientation) or record why no further tissue may be taken.
  Arms: Device

SUMMARY:
This is a multi-center, randomized, two-arm study designed to measure the effectiveness of the SELENE system in reducing the number of unaddressed positive margins in breast lumpectomy procedures when used in addition to standard intraoperative margin assessment.

ELIGIBILITY:
Inclusion Criteria:

* Female
* Age 18 years or older
* Patients undergoing elective breast conservation surgery for the treatment of Stage 0-III invasive ductal and/or ductal carcinoma in situ
* May include subjects treated with neo-adjuvant therapy (endocrine and/or chemotherapeutic), but not required for study inclusion
* Ability to understand and the willingness to sign a written informed consent document

Exclusion Criteria:

* Male
* Metastatic cancer (Stage IV)
* Lobular carcinoma as primary diagnosis
* Previous ipsilateral breast surgery for benign or malignant disease within two years (this includes implants and breast augmentation)
* Subjects with multi-centric disease (histologically diagnosed cancer in two different quadrants of the breast), unless resected in a single specimen
* Subjects with bilateral disease (diagnosed cancer in both breasts)
* Participating in any other investigational margin assessment study which can influence collection of valid data under this study
* Use of cryo-assisted localization
* Currently lactating
* Current pregnancy
* Subjects for whom the specimen margins have been destroyed, damaged, or are otherwise not intact prior to imaging (device arm only) imaging

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 482 (Actual)
Dates: Start 2021-12-01 (Actual); Primary Completion 2024-09-23 (Actual); Study Completion 2024-10-21 (Actual)

PRIMARY OUTCOMES:
The occurrence of at least one unaddressed positive margin for a subject. | Pathology report finalization date, usually 3-7 days post-surgery
  Within-subject comparison of the occurrence of subjects with at least one positive margin.

SECONDARY OUTCOMES:
The number of unaddressed positive margins per subject. | Pathology report finalization date, usually 3-7 days post-surgery
  The average number of unaddressed positive margins per subject.
False Positive Shaves Per Subject | Pathology report finalization date, usually 3-7 days post-surgery
  The number of false-positive shaves per subject with use of SELENE.
Margin-level effectiveness (National Guidelines) | Pathology report finalization date, usually 3-7 days post-surgery
  Margin-level effectiveness of SELENE based on recorded clinical decisions with "ground truth" determined based on National Comprehensive Cancer Network (NCCN), Society of Surgical Oncology (SSO), and the American Society for Radiation Oncology (ASRO) Guidelines (device arm Part B only- all margins)
Margin-level effectiveness (Histopathology) | Pathology report finalization date, usually 3-7 days post-surgery
  Margin-level effectiveness of SELENE based on recorded clinical decisions with "ground truth" determined based on histopathological presence of disease at 2 mm or less based on visible tissue depth using OCT (device arm Part B only- all margins)

OTHER OUTCOMES:
Safety Outcome - Adverse Events | Throughout study duration
  Assessed by recording all adverse events for the duration of the study and then analyzing by seriousness, severity, and device/SELENE procedure-relatedness.
Safety Outcome - Patient Reported Outcome | Prior to index surgical visit and between 4-12 weeks post-surgical date
  Pre- and Post-operative satisfaction with breasts using the Satisfaction with Breasts subscale score of the BCT module of the patient-reported outcomes measurement instrument BREAST-Q.

CONTACTS AND LOCATIONS:
Locations (10):
- United States (10):
  - Baptist MD Anderson Cancer Center, Jacksonville, Florida
  - Mayo Clinic, Jacksonville, Florida
  - Moffitt Cancer Center & Research Institute, Tampa, Florida
  - Holy Redeemer, Meadowbrook, Pennsylvania
  - West Cancer Center & Research Institute, Germantown, Tennessee
  - Medical City Dallas, Dallas, Texas
  - Baylor College of Medicine, Houston, Texas
  - Methodist Healthcare of San Antonio, San Antonio, Texas
  - University of Washington, Seattle, Washington
  - University of Wisconsin, Madison, Wisconsin

IPD SHARING:
Plan to Share IPD: No